CLINICAL TRIAL: NCT05526651
Title: Improvement of Urinary Retention Symptoms After Vaginal Delivery With Electroacupuncture Therapy
Brief Title: Improvement of Urinary Retention Symptoms With Electroacupuncture Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Ayu Permata Sari, Medical doctor, student of medical acupuncture specialist program, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-08-0889
Record Dates: First submitted 2022-08-28; First posted 2022-09-02 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Urinary Retention
Keywords: Urinary Retention; Postpartum urinary retention; electroacupuncture; vaginal delivery; acupuncture
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Study divided into 2 arms, true electroacupuncture group and sham electroacupuncture group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True electroacupuncture group (Experimental): the investigators use stainless steel acupuncture needle, disposable : Huanqiu® 0.25 x 0.40 mm Electroacupuncture device : Hwato-SDZ V®, continuous wave, 2 Hz, for 30 minutes
  Interventions: Other: true electroacupuncture
- sham electroacupuncture group (Sham Comparator): the investigators use the same device like true electroacupuncture group, but the acupuncture needle not puncture on the skin and only attached.
  electroacupuncture device, with no electrical stimulation
  Interventions: Other: sham electroacupuncture

INTERVENTIONS:
Other: true electroacupuncture — the investigators use stainless steel acupuncture needle, disposable : Huanqiu® 0.25 x 0.40 mm Electroacupuncture device : Hwato-SDZ V®, continuous wave, 2 Hz, for 30 minutes
  Arms: True electroacupuncture group
Other: sham electroacupuncture — the investigators use the same device like true electroacupuncture group, but the acupuncture needle not puncture on the skin and only attached.
  electroacupuncture device, with no electrical stimulation
  Arms: sham electroacupuncture group

SUMMARY:
Postpartum urinary retention (PPUR) can occur in women who deliver vaginally. The incidence of this occurrence varies from 1.7 - 17.9%, this different variation due to different definitions of PPUR and the methods used to measure it. There are 2 categories of RUPP, namely covert and overt, in overt PPUR the prevalence ranges from 0.3 to 4.7%, while covert PPUR can reach up to 45%. In Indonesia alone, the incidence of PPUR is around 14.8%3, where vaginal PPUR is around 70% more higher than sectio caesarean patients. A study conducted at the RSCM in 2009 by Yustini, et al stated that the incidence of PPUR was 9-14%, and if the delivery was using forceps it would increase to 38%. Other studies conducted by Suskhan at the RSCM in 2015, it was stated that the incidence of urinary retention was 13.6% of 500 research subjects. Another study conducted by Chen, et al in 2020 in China, stated that the most common cause of urinary retention in hospitals was surgery. gynecological cases, which is 69% while for obstetric cases by 18.6% where the main cause of this retention is due to vaginal delivery. The high number of PPUR can increase the incidence of postpartum hemorrhage, urinary tract infections, mental fatigue during the puerperium and result in delays in breastfeeding. Bladder catheterization which is one of the treatments for PPUR is also closely related to the risk the occurrence of morbidity and complications, where 17.5% of urinary tract infections are infections obtained from hospitals or HAIs (Healthcare Associated Infections) and 80% of these infections are caused by the installation of urethral catheters, especially the installation of urethral catheters in the ER which is carried out without clear indications such as described in a study conducted by Gokula et al in Michigan in 2007.

According to Sudhakaran, symptomatic RUPP (overt) is defined as the absence of a spontaneous voiding process or the inability to urinate since 6 hours after vaginal delivery or 6 hours after catheter removal after caesarean section. Asymptomatic (covert) PPUR is defined as a post-void residual volume (PVRV) 200 ml after the first spontaneous urination as measured by ultrasound or catheter, which indicates incomplete voiding.6 Asymptomatic PPUR may occur due to reduced sensation and contractility that occurs as a result of trauma from the innervation to the bladder. Symptoms of this RUPP according to Suskhan are unexplained urination, prolonged urination, more frequent urination, inability to urinate, feeling of full bladder and abdominal distension. The presence of the above symptoms will cause the bladder to enlarge during a physical examination of the abdomen.

Acupuncture as a non-medical therapy has been widely used both in China and in other countries, especially to treat pain and neurological disorders. Urination is a neural reflex activity. Acupuncture points that correspond to the innervation of the bladder can stimulate conduction of parasympathetic nerve impulses, resulting in bladder detrusor contraction, increased intravesical pressure and relaxation of the internal sphincter. Thus, acupuncture can regulate bladder function in the process of urination.

Based on the study of Zhao, et al, it was stated that electroacupuncture can stimulate afferent and efferent nerves in the pelvic cavity of rats, increase detrusor contraction and encourage urination. Other studies have shown that electroacupuncture can also reduce the myoelectric activity of abnormal contraction of the external urethral sphincter during urination, reduce resistance during urination, improve coordination between the bladder detrusor and urethral sphincter and reduce residual urine volume. As for the side effects caused by acupuncture based on a systematic study conducted almost none.

Based on the description above, acupuncture can be considered as a supportive therapy that can overcome the problem of PPUR with minimal side effects to prevent worsening of the condition. In this study, researchers wanted to determine the effectiveness of acupuncture interventions using electroacupuncture modalities to accelerate urination after delivery and reduce residual urine volume in patients after vaginal delivery with electroacupuncture intervention for 30 minutes / session, 2 sessions in 1 x 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* subject who had urinary retention 6 hours after vaginal delivery and the residual urine volume 500 - 1000 mL
* female 20 - 40 years old
* pregnancy > 34 weeks and baby's weight > 2000 gr
* agree to participate in this study and sign the inform consent

Exclusion Criteria:

* patient who had emergency situation, such as bleeding or unstable hemodynamic
* using pace maker
* had cardiac arrhythmia
* patient had disease that make them using the catheter (such as chronic kidney disease)
* allergy to stainless steel
* scar in the acupuncture point locations
* using prothesis
* had intrathecal labour analgesia (ILA)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
residual urine volume after electroacupuncture therapy and catheter removal | 6 hours
  after 24 hours using catheter, it will be remove. 6 hours after catheter removal, the investigators will check how much the residual urine volume in the bladder

SECONDARY OUTCOMES:
first time micturation | 6 hours
  after 24 hours using catheter, it will be remove. anytime after the removal if participants going to first micturition, the investigators will collect the data

CONTACTS AND LOCATIONS:
Locations (1):
- Koja Regional Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided